CLINICAL TRIAL: NCT03738436
Title: The Effects of Adding Modified Visual Feedback Training in Physical Therapy Protocol Following Anterior Cruciate Ligament Reconstruction
Brief Title: Adding Modified Visual Feedback Training in Patients Following ACL Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsiu-Chen Lin, Associate Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC3-124
Record Dates: First submitted 2018-10-31; First posted 2018-11-13 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Visual feedback; Proprioception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional neuromuscular training, NMT (Active Comparator): Eight-week physical therapy program consisted of neuromuscular training (NMT) starting from 4 weeks post-surgery. The NMT program includes re-position exercise, strengthening, stretching, landing and balance training.
  Interventions: Other: Physical therapy traditional neuromuscular training, NMT
- modified visual feedback, MVF (Experimental): Starting from 4 weeks post-surgery, eight-week physical therapy program consisted of traditional neuromuscular training (as in NMT group), but with modified visual feedback by eyes closed, reduced lighting or wearing strobe goggles.
  Interventions: Other: Physical therapy modified visual feedback, MVF

INTERVENTIONS:
Other: Physical therapy traditional neuromuscular training, NMT — The NMT program includes re-position exercise using Swiss ball roll squat, strengthening and stretching exercises in various positions or combined using Swiss ball, Thera-Band or suspension system (Redcord), balance exercise on wobble board, proper landing strategy practices, and etc.
  Other Names: The neuromuscular training (NMT) program
  Arms: traditional neuromuscular training, NMT
Other: Physical therapy modified visual feedback, MVF — traditional neuromuscular training (as in NMT group), but with modified visual feedback by eyes closed, reduced lighting or wearing strobe goggles
  Arms: modified visual feedback, MVF

SUMMARY:
The current treatment for the ACL-injured patients usually emphasize on the movement quality through neuromuscular training. The purpose of this study is to (1) design a modified visual feedback training program and (2) investigate the effects of the modified visual feedback training on the movement control in the ACL-reconstructed (ACL-R) patients. Forty unilateral ACL-R male patients will be enrolled voluntarily, who will be randomly allocated into the traditional neuromuscular training (NMT) or the modified visual feedback (MVF) group. The investigators hypothesize that this MVF training program will have better potential to improve their post-injury movement dysfunction.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) rupture is a common sport-related injury that needs surgical reconstruction to restore a better knee function. This ligament accommodates plenty of crucial sensory nerve endings providing proprioceptive information to central nerve system (CNS) for the knee movement control. Recent studies have found that the patients will increase utilization of the visual processing for movement control, concurrent with the depression of the proprioceptive information after the ACL injury. In addition, the loss of proprioception information will result in motor impairment when disrupting vision during more demanding physical activities, such as pivoting, accelerating, decelerating, and landing maneuver. It is obvious that this motor control deficit may increase the re-injury risk during multitasking situations common in functional movements or sports participation. The current treatment for the ACL-injured patients usually emphasize on the movement quality through neuromuscular training, but seldom adding the alteration of the sensory processing. Some patients still have been forced to lower their activity level or ended their career in sports due to the remained motor control problems after rehabilitation. Therefore, the purpose of this study is to (1) design a modified visual feedback training program and (2) investigate the effects of the modified visual feedback training on the movement control in the ACL-reconstructed (ACL-R) patients. Forty unilateral ACL-R male patients will be enrolled voluntarily from local hospitals to participate in this study. Each participant will be randomly allocated into the traditional neuromuscular training (NMT) or the modified visual feedback (MVF) group. The training program will start at the forth week after the ACL reconstruction and last for eight weeks. The hypothesis of this study is that the MVF training program will have better potential to improve their post-injury movement dysfunction and thus may decrease the re-injury risk in ever-changing environment. Therefore, it may provide assistance for the patients to build both physical and neurocognitive capabilities for returning to sport.

ELIGIBILITY:
Inclusion Criteria:

* unilateral ACL injury male patients aged from 20~45 years old
* arthroscopic assisted ACL reconstruction with autologous patellar tendon or hamstring tendon graft
* no other knee injury
* no limited range of motion at the hip or ankle joints

Exclusion Criteria:

* injuries in the other knee joint
* previous injuries in the ipsilateral hip or ankle joints
* neurological disease that affects his motor function

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-02 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Position sense (Proprioception) of the knee joints | Change from post-operative 4 weeks to post-operative 13 weeks
  It will be performed on a isokinetic machine (Biodex System 3) to obtain the error angles (degrees) in the test of the joint position reproduction (JPR)
Movement sense (Proprioception) of the knee joints | Change from post-operative 4 weeks to post-operative 13 weeks
  It will be performed on a isokinetic machine (Biodex System 3) to obtain the angles (in degrees) in the test of threshold to detection of passive motion (TTDPM)
Maximal muscle strength | Change from post-operative 4 weeks to post-operative 13 weeks
  Maximal isometric strength (in torque, Nm) of knee extensor & flexor will be tested on the isokinetic machine (Biodex System 3)
Balance Test | Change from post-operative 4 weeks to post-operative 13 weeks
  Y Balance Test (YBT) - The test requires the participant to balance on one leg while reaching as far as possible with the other leg in three separate directions: anterior, posterolateral, and posteromedial. The composite score (in percentage, %) of summarized reaching distances, each divided by leg length first, in three directions will be recorded.

SECONDARY OUTCOMES:
Functional outcome questionnaire | Change from post-operative 4 weeks to post-operative 13 weeks
  A self-administered 14-item questionnaire - Knee Outcome Survey - Activities of Daily Living Scale (KOS-ADLS) will be used to evaluate the symptom-related (6 items) and specific functional limitations during ADL (8 items). The responses are graded on a 6-point Likert scale (0 to 5 points), with 5 indicating no symptom or limitation and 0 indicating the severest limitation. The total score is 70 points, and then will be transformed to a 0- to 100-point scale (percentage of disability).

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chen Lin, PhD, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No